CLINICAL TRIAL: NCT01465152
Title: Multicentre, Randomised, Comparative, Open, Three Armed Parallel Group Study on the Use of Metformin, Repaglinide or the Combination of Both in Type 2 Diabetic Patients After Failure of Dietary Measures
Brief Title: Comparison of Metformin, Repaglinide or the Combination of Both in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-1411
Record Dates: First submitted 2011-10-31; First posted 2011-11-04 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Metformin; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Met (Experimental)
  Interventions: Drug: metformin
- Rep (Active Comparator)
  Interventions: Drug: repaglinide
- Met+Rep (Active Comparator)
  Interventions: Drug: metformin; Drug: repaglinide

INTERVENTIONS:
Drug: metformin — Adminstered orally during the three main meals for 24 weeks
  Arms: Met; Met+Rep
Drug: repaglinide — Administered orally before the three main meals for 24 weeks
  Arms: Met+Rep; Rep

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the efficacy of metformin and repaglinide used alone or combined administered as initial treatment in subjects with type 2 diabetes in which diet and exercise have failed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Treated by diet for at least 3 months
* Never treated with hypoglycaemic drugs
* HbA1c (glycaemic haemoglobin A1c) on inclusion time superior to 6.5%

Exclusion Criteria:

* Very symptomatic diabetes
* Advanced vascular complications
* Manifest renal failure
* Manifest hepatic disease
* Pregnancy, breast feeding or intention to become pregnant or if it is considered that the patient is not using adequate contraceptive measures. Adequate contraceptive measures are considered to be an intrauterine device, oral contraceptives and barrier methods

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2002-03-06 (Actual); Primary Completion 2004-10-21 (Actual); Study Completion 2004-10-21 (Actual)

PRIMARY OUTCOMES:
Change of % HbA1c (glycosylated haemoglobin) in blood

SECONDARY OUTCOMES:
Change of the mean body mass index calculated as weight in kilograms divided by the square of height in metres
Incidence of clinical and/or biochemistry hypoglycaemia episodes
Incidence of adverse events
Presence of laboratory abnormalities in routine blood analyses
Change of the blood pressure and/or heart rate
Treatment compliance

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (15):
- Spain (15):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Benamargosa
  - Novo Nordisk Investigational Site, Burlata
  - Novo Nordisk Investigational Site, Camas
  - Novo Nordisk Investigational Site, Fuenlabrada
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Lugo
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Portugalete
  - Novo Nordisk Investigational Site, San Adria Del Besos
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Tegueste
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Zaragoza

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com